CLINICAL TRIAL: NCT02604602
Title: Peripartal Concentration of Coagulation Factors and Postpartum Hemorrhage
Brief Title: Coagulation Factors and Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0011
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Postpartum Hemorrhage
Keywords: PPH
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PPH
  Interventions: Other: blood exam
- non-PPH
  Interventions: Other: blood exam

INTERVENTIONS:
Other: blood exam — laboratory test

SUMMARY:
Objective is to analyze a possible association of coagulation factors peripartal with the occurrence of postpartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women > 22 weeks of gestation

Exclusion Criteria:

* age < 18 years, no informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women before delivery
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-10; Primary Completion 2018-11 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
occurrence of PPH | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Haslinger, M.D., Principal Investigator — Division of Obstetrics, University Hospital of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland